CLINICAL TRIAL: NCT04053972
Title: The Impact on Recurrence Risk of Adjuvant Lenvatinib for Patients With Hepatocellular Carcinoma And Microvascular Invasion (MVI) After Hepatectomy : A Random, Controlled, Stage III Clinical Trial.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rong-ping Guo, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2019-042-01
Record Dates: First submitted 2019-08-10; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): adjuvant lenvatinib
  Interventions: Drug: Lenvatinib
- control group (No Intervention): no intervention

INTERVENTIONS:
Drug: Lenvatinib — oral lenvatinib after hepatectomy
  Arms: treatment group

SUMMARY:
To compare The Impact on Recurrence Risk of Adjuvant Lenvatinib for Patients With Hepatocellular Carcinoma And Microvascular Invasion (MVI) After Hepatectomy.

ELIGIBILITY:
No

Criteria:

Inclusion Criteria:

older than 18 years old and younger than 75 years; ECOG PS<3; proven hepatocellular carcinoma with MVI according pathological examination; not previous treated for tumor; tumor was removed in operation; no recurrence occurence at 4 to 7 weeks after surgery; the lab test could meet: neutrophil count≥1.5×109/L; hemoglobin≥80g/L; platelet count≥60×109/L; serum albumin≥28g/L; total bilirubin<3-times upper limit of normal; ALT<5-times upper limit of normal; AST<5-times upper limit of normal; serum creatine<1.5-times upper limit of normal; PT≤upper limit of normal plus 6 seconds; INR≤2.3; sign up consent; unrolled by other clinical trials about hepatocellular carcinoma.

Exclusion Criteria:

cannot tolerate lenvatinib; CNS or bone metastasis exits; known history of other malignancy; be allergic to related drugs; underwent organ transplantation before; be treated before (interferon included); known history of HIV infection; known history of drug or alcohol abuse; have GI hemorreage or cardiac/brain vascular events within 30 days; pregnancy;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
RFS | From date of randomization until the date of recurrence, assessed up to 60 months
  recurrence-free survival

SECONDARY OUTCOMES:
OS | From date of randomization until the date of death from any cause, assessed up to 60 months
  overall survival
recurrence rate | 1 year, 2 year, 3 year, 5 year after surgery
  recurrence rate

CONTACTS AND LOCATIONS:
Locations (1):
- SUN YAT-SEN University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided